CLINICAL TRIAL: NCT00617292
Title: Long-Term Outcome in Offspring and Mothers of Dexamethasone-Treated Pregnancies at Risk for Classical Congenital Adrenal Hyperplasia Owing to 21-Hydroxylase Deficiency
Brief Title: Determining the Long-Term Effects of Prenatal Dexamethasone Treatment in Children With 21-Hydroxylase Deficiency and Their Mothers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Office of Rare Diseases (ORD) (NIH)
Responsible Party: Maria I. New, MD, Mount Sinai School of Medicine
Other Study IDs: RDCRN 5610
Record Dates: First submitted 2008-01-31; First posted 2008-02-18 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Adrenal Hyperplasia, Congenital
Keywords: 21-hydroxylase deficiency; 21OHD; CAH
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Category 1, Group 1: Children who have 21OHD and received prenatal dexamethasone treatment
- Category 1, Group 2: Children who have 21OHD and did not receive prenatal dexamethasone treatment (control)
- Category 2: Mothers of children who received prenatal dexamethasone treatment

SUMMARY:
Congenital adrenal hyperplasia (CAH) is a genetic disorder that affects the amount of steroids that the body forms. The most common form of CAH is 21-hydroxylase deficiency (21OHD), which leads to cortisol deficiency and causes the development of mature masculine characteristics in newborn, prepubescent, and grown females, and prepubescent males. Prenatal treatment with dexamethasone, a corticosteroid, has been shown to reduce the masculinization of genitalia. However, the long-term effects of dexamethasone on the children who received it as fetuses and on mothers who were exposed to it while they were pregnant have not been determined. This study will investigate potential long-term adverse side effects of prenatal dexamethasone treatment in children and young adults who received dexamethasone as fetuses and their mothers who were exposed to it during pregnancy.

DETAILED DESCRIPTION:
CAH is a genetic steroidogenesis disorder. The most common form, 21OHD, leads to cortisol deficiency and, in turn, an excess of androgen, a hormone that promotes the development and maintenance of male sex characteristics. As a result of this androgen excess, prepubescent males and newborn, prepubescent, and grown females exhibit mature masculine characteristics. Prenatal treatment with dexamethasone, a corticosteroid that decreases androgen levels, has been shown to prevent the development of abnormal genitalia in female infants. The long-term effects of this treatment, however, have not been evaluated. This study will determine whether prenatal dexamethasone treatment causes any long-term side effects by examining children and young adults who received dexamethasone as fetuses and their mothers, who were exposed to dexamethasone while pregnant.

This study has three parts. In Part 1 of the study, participants will provide written consent for release of their medical records from their physicians. Participants' physicians will then complete a medical form and/or provide copies of selected medical records for each participant. Parts 2 and 3 can be completed in 1 day. In Part 2 of the study, participants will complete questionnaires in their homes. Participants will answer questions about the following experiences: medical procedures, such as hormone treatment and genital surgery; education; work; hobbies; play activities and chores during childhood; identification with the male or female gender; relationships with parents; interest in being a parent; and overall adjustment. Part 3 of the study will consist of neuropsychological testing at the study site. This testing will focus on memory, attention, and overall cognitive abilities.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* English-speaking
* Has undergone DNA testing for mutations in the CYP21A2 gene

For children who received prenatal dexamethasone treatment:

* Genetic confirmation of 21OHD diagnosis
* Received full or partial prenatal dexamethasone treatment

For children in the control group:

* Did not receive prenatal dexamethasone treatment

For mothers:

* History of at-risk pregnancy for a fetus affected with 21OHD
* Genetic confirmation of child's diagnosis

Exclusion Criteria:

* Any mental disorder that could prevent understanding of study materials
* Current or past steroid use for reasons other than CAH (i.e., asthma, lupus, rheumatoid arthritis)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study will include children who received prenatal dexamethasone treatment as fetuses and their mothers.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypertension and obesity | Throughout the study
"Normal" masculinization of unaffected females treated prenatally with dexamethasone | Throughout the study
Normal masculinization of male fetuses partially treated prenatally with dexamethasone | Throughout the study
Memory-related cognitive function | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Maria I. New, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- University of Sao Paolo, São Paulo, São Paulo, Brazil
- University of Lyon, Lyon, France